CLINICAL TRIAL: NCT04239027
Title: A One-year, Single-arm, Open-label, Multicenter Study Assessing the Anatomic Outcomes of Brolucizumab Assessed by OCT-A in Adult Patients With Neovascular Age Related Macular Degeneration
Brief Title: A Study to Assess the Effects of Brolucizumab in Adult Patients With Neovascular Age Related Macular Degeneration
Acronym: OCTOPUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRTH258AFR01; 2019-003338-17 (EudraCT Number)
Record Dates: First submitted 2020-01-21; First posted 2020-01-23 (Actual); Results first posted 2024-06-04 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Neovascular Age Related Macular Degeneration
Keywords: age-related macular degeneration, wetAMD, nAMD, neovascular, choroidal neovascularization, CNV, OCT-angiography
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — brolucizumab

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RTH258/Brolucizumab (Experimental): This is a single-arm study in which all patients will be treated with brolucizumab 6mg: 3 loading injections (at Screening/Baseline, Week 4 and Week 8), followed by maintenance treatment from Week 16/Week 20 up to Week 40/Week 44.
  Interventions: Drug: RTH258/Brolucizumab

INTERVENTIONS:
Drug: RTH258/Brolucizumab — Brolucizumab is a new generation of anti-VEGF (vascular endothelial growth factor). All patients were treated with brolucizumab 6mg: 3 loading injections (at Screening/Baseline, Week 4 and Week 8), followed by maintenance treatment every 8 weeks (Q8W) or every 12 weeks (Q12W) depending on disease activity from Week 16/Week20 to Week 40/Week 44.
  Brolucizumab was administered by an intravitreal (IVT) injection to the study. eye.

SUMMARY:
Neovascular age-related macular degeneration (nAMD) is characterized by the presence of choroidal neovascularization (CNV). Choroidal neovascularization consists of abnormal blood vessels originating from the choroid and can lead to hemorrhage, fluid exudation, and fibrosis, resulting in photoreceptor damage and vision loss.

The safety and efficacy of brolucizumab has been demonstrated in 2 randomized, multicenter, double-masked, active controlled Phase 3 studies in nAMD patients (RTH258-C001 and RTH258-C002). Anatomical changes were evaluated in these studies using spectral domain optical coherence tomography (SD-OCT), which relied on indirect parameters for the diagnosis of active CNV. The OCT-angiography (OCT A) that directly visualize retinal circulation and image CNV and vascular diseases of the retina was not included in previous brolucizumab studies.

This single-arm, open-label, multicenter study was performed to evaluate the efficacy and safety of brolucizumab 6 mg in patients with nAMD.

OCT-A was used in this study to assess the morphological response of patients to brolucizumab in terms of percentage change in CNV lesion area in the short term (i.e. at Week 12) and in the long term (i.e. at Week 48), as well as changes in other OCT-A features up to Week 48.

DETAILED DESCRIPTION:
This was a prospective, single-arm, open-label, multicenter study to evaluate the efficacy and safety of brolucizumab 6 mg in patients with neovascular age-related macular degeneration (nAMD). Patients were required to attend 6 mandatory study visits: Screening/Baseline Visit (Day 1), Week 4, Week 8, Week 12, Week 16 and Week 48 visits. The timing of the interim visits between Week 16 and Week 48 depended on the patient's injection regimen, i.e. every 12 weeks (q12w) or every 8 weeks (q8w). Patients who consented and met all the inclusion and none of the exclusion criteria were screened to evaluate eligibility. After confirmation of eligibility, patients were included and treated with brolucizumab 6 mg. The maximum study duration for 1 patient was 48 weeks, including Screening. There were 2 periods in this study:

* Open-label treatment period: from Screening/Baseline (Day 1) to Week 40/Week 44 (depending on assigned regimen)
* Follow-up period: Week 40/Week 44 to Week 48

A Safety Review Committee (SRC) was established for this study to provide an independent, systematic, standardized and unbiased assessment of the review of intraocular inflammation (IOI), retinal vasculitis (RV) and/or retinal vascular occlusion (RO).

ELIGIBILITY:
INCLUSION Criteria:

1. Patients must provide written informed consent before any study related procedures are performed.
2. Patients must be 50 years of age or older at Screening/Baseline.

   Study eye:
3. Active CNV lesions secondary to AMD that affect the central subfield, including retinal angiomatous proliferation (RAP) with a CNV component, confirmed by presence of active leakage from CNV seen by fluorescein angiography and sequellae of CNV, e.g. pigment epithelial detachment (PED), subretinal hemorrhage or sub-retinal pigment epithelium (sub-RPE) hemorrhage, blocked fluorescence, macular edema.
4. Intra- and/or subretinal fluid affecting the central subfield of the study eye at Screening/Baseline.
5. BCVA between 83 and 23 letters, inclusive, in the study eye at Screening/Baseline using early treatment diabetic retinopathy study (ETDRS) at an initial testing distance of 4 meters.

EXCLUSION Criteria:

Ocular conditions:

1. Any active intraocular or periocular infection or active intraocular inflammation (e.g. infectious conjunctivitis, keratitis, scleritis, endophthalmitis, infectious blepharitis) in either eye at Screening/Baseline.
2. Presence of amblyopia, amaurosis or ocular disorders in the fellow eye with BCVA < 35 ETDRS letters at Screening (except when due to conditions whose surgery may improve visual acuity, e.g. cataract).
3. Medical history of intraocular inflammation and/or retinal vascular occlusion within 12 months prior to Screening/Baseline.

   Study eye:
4. Poor quality of OCT-A and SD-OCT images at Screening/Baseline.
5. Atrophy or fibrosis involving the center of the fovea in the study eye, as assessed by color fundus photography and fundus autofluorescence (FAF) at Screening/Baseline.
6. The total area of fibrosis or subretinal blood affecting the foveal center point comprising ≥ 50% of the lesion area in the study eye at Screening/Baseline.
7. Concomitant conditions or ocular disorders in the study eye, including retinal diseases other than nAMD, that, in the judgment of the investigator, could require medical or surgical intervention during the course of the study to prevent or treat visual loss that might result from that condition, or that limits the potential to gain visual acuity upon treatment with the investigational product.
8. Structural damage within 0.5 disc diameter of the center of the macula in the study eye, e.g. vitreomacular traction, epiretinal membrane, retinal pigment epithelium (RPE) rip/tear scar, laser burn, at the time of Screening that in the investigator's opinion could preclude visual function improvement with treatment.
9. Current vitreous hemorrhage or history of vitreous hemorrhage in the study eye within 4 weeks prior to Screening/Baseline.
10. Uncontrolled glaucoma in the study eye defined as IOP > 25 mmHg on medication or according to the investigator's judgment at Screening/Baseline.
11. Aphakia and/or absence of the posterior capsule in the study eye at Screening/Baseline.

    Ocular treatments (study eye):
12. Patient has received any approved or investigational treatment for nAMD (other than vitamin supplements) in the study eye at any time.
13. Intraocular or periocular use of corticosteroids in the study eye during the 6-month period prior to Screening/Baseline.
14. Previous penetrating keratoplasty or vitrectomy at any time prior to Screening/Baseline.
15. History or evidence of the following in the study eye within the 90-day period prior to Screening/Baseline:

    * Intraocular or refractive surgery.
    * Previous panretinal photocoagulation.
    * Previous submacular surgery, other surgical intervention or laser treatment for nAMD including photodynamic therapy (PDT).

    Systemic conditions or treatments:
16. End stage renal disease requiring dialysis or renal transplant.
17. Systemic medications known to be toxic to the lens, retina or optic nerve (e.g. deferoxamine, chloroquine/hydroxychloroquine, tamoxifen, phenothiazines and ethambutol) used during the 6-month period prior to Screening/Baseline except temporary use for COVID-19 treatment.
18. Participation in an investigational drug, biologic, or device study within 30 days or the duration of 5 half-lives of the investigational product (whichever is longer) prior to Screening/Baseline. Note: observational clinical studies solely involving over-the-counter vitamins, supplements, or diets are not exclusionary.
19. Systemic anti-VEGF therapy at any time.
20. Stroke or myocardial infarction in the 6-month period prior to Screening/Baseline.
21. Uncontrolled blood pressure defined as a systolic value ≥ 160 mmHg or diastolic value ≥ 100 mmHg at Screening/Baseline. (In case there is an elevated blood pressure measurement, it should be repeated after 20 minutes. If the repeat measurement is elevated, then the patient is not eligible to be enrolled into the study).
22. History of a medical condition (disease, metabolic dysfunction with exception of type 1 or 2 diabetes mellitus, physical examination finding, or clinical laboratory finding) that, in the judgment of the investigator, would preclude scheduled study visits, completion of the study, or a safe administration of investigational product.
23. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
24. History of hypersensitivity to any component of the test article, control article, or clinically relevant sensitivity to fluorescein dye, as assessed by the investigator.

    Other:
25. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) pregnancy test.
26. Women of childbearing potential, defined as all women less than 1 year postmenopausal or less than 6 weeks since sterilization at Screening/Baseline Women are considered post-menopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks before taking study treatment. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of childbearing potential.
27. Patients mentioned in Articles L.1121-5 to L.1121-8 and L.1122-1-2 of the Code de Santé Publique (e.g. minors, protected adults, etc.)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (37):
- France (37):
  - Novartis Investigative Site, Nice, Cedex1
  - Novartis Investigative Site, Rennes, FRA
  - Novartis Investigative Site, Saint-Cyr-sur-Loire, Indre Et Loire
  - Novartis Investigative Site, Lyon, Rhone
  - Novartis Investigative Site, Bobigny, Seine Saint Denis
  - Novartis Investigative Site, Aix-en-Provence
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Boulogne-sur-Mer
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Floirac
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, La Rochelle
  - Novartis Investigative Site, Lagord
  - Novartis Investigative Site, Le Chesnay
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montargis
  - Novartis Investigative Site, Montauban
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Mulhouse
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Perpignan
  - Novartis Investigative Site, Plérin
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Royan
  - Novartis Investigative Site, Rueil-Malmaison
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Saint-Martin-des-Champs
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://clinicalstudydatarequest.com/Default.aspx

REFERENCES:
- [Derived] Bodaghi B, Souied EH, Tadayoni R, Weber M, Ponthieux A, Kodjikian L. Detection and Management of Intraocular Inflammation after Brolucizumab Treatment for Neovascular Age-Related Macular Degeneration. Ophthalmol Retina. 2023 Oct;7(10):879-891. doi: 10.1016/j.oret.2023.06.009. Epub 2023 Jun 19. PMID 37343623
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1874

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 210 adult patients were treated at 40 centers in France. The maximum study duration for 1 patient was 48 weeks.
Pre-assignment Details: The Screening/Baseline visit were performed on the same Visit (Day 1). The first dose of study treatment was also administered on Day 1.
Groups:
- RTH258/Brolucizumab: This is a single-arm study in which all patients were treated with brolucizumab 6mg: 3 loading injections (at Screening/Baseline, Week 4 and Week 8), followed by maintenance treatment from Week 16/Week 20 up to Week 40/Week 44.
Period: Overall Study
Arm/Group | RTH258/Brolucizumab
Started | 210
Completed | 184
Not Completed | 26
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 9
Not completed — Death | 1
Not completed — Physician Decision | 9
Not completed — Lost to Follow-up | 2
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 210
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.8 (7.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129
  Male | 81
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Choroidal Neovascularization (CNV) Lesion Area Measured by Optical Coherence Tomography-Angiograph (OCT-A) From Baseline to Week 12
Description: OCT-A is a dye-less angiographic procedure based on split-spectrum-decorrelation-amplitude angiography.
  It enables the capture of scattered intra-vessel particles (mainly erythrocyte cells) at all levels of the retinal and inner-choroidal vasculature, thus providing 3-D imaging of the retinal circulation.
  The literature suggests that OCT-A is a good marker for assessing anti-VEGF therapeutic response, especially lesion size.
  Inter-Quartile Range = q1 - q3.
Time Frame: Baseline, Week 12
Population: Participants in the Full Analysis Set (FAS) with a valid value for the outcome measure. The FAS is comprised of all treated patients.
  Due to ungradable images and other reasons, only 138 patients were evaluable at Week 12 for choroidal neovascularization (CNV) lesion area by optical coherence tomography-angiography (OCT-A) in nAMD. This sample size of 138 patients was reassessed and shown to be valid for analysis of the primary efficacy endpoint.
Measure: Median (Inter-Quartile Range); unit: % change from baseline
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 138
% change from baseline | -79.29 [-100.00 to -11.19]

2. Secondary Outcome: Percentage Change in Choroidal Neovascularization (CNV) Lesion Area Measured by Optical Coherence Tomography-Angiograph (OCT-A) From Baseline to Week 48
Description: OCT-A is a dye-less angiographic procedure based on split-spectrum-decorrelation-amplitude angiography.
  It enables the capture of scattered intra-vessel particles (mainly erythrocyte cells) at all levels of the retinal and inner-choroidal vasculature, thus providing 3-D imaging of the retinal circulation.
  The literature suggests that OCT-A is a good marker for assessing anti-VEGF therapeutic response, especially lesion size.
Time Frame: Baseline, Weeks 4, 8, 48
Population: Participants in the Full Analysis Set (FAS) with a valid value for the outcome measure at baseline and at each timepoint. The FAS comprised all patients to whom study treatment had been assigned and who received at least one IVT injection of study treatment.
Measure: Median (Inter-Quartile Range); unit: % change from baseline
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 124
% change from baseline
  Week 4 (n=124) | -59.03 [-100.00 to -6.34]
  Week 8 (n=109): number analyzed (Participants) | 109
  Week 8 (n=109) | -53.41 [-100.00 to -0.67]
  Week 48 (n=117): number analyzed (Participants) | 117
  Week 48 (n=117) | -68.50 [-100.00 to -1.40]

3. Secondary Outcome: Change in Choroidal Neovascularization (CNV) Lesion Area Measured by Optical Coherence Tomography-Angiograph (OCT-A) From Baseline to Week 48
Description: as for outcome 2
Time Frame: Baseline, Weeks 4, 8, 12, 48
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: square millimeters
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 140
square millimeters
  Week 4 (n=126): number analyzed (Participants) | 126
  Week 4 (n=126) | -0.09 [-0.34 to -0.00]
  Week 8 (n=111): number analyzed (Participants) | 111
  Week 8 (n=111) | -0.12 [-0.47 to 0.00]
  Week 12 (n=140) | -0.14 [-0.50 to -0.01]
  Week 48 (n=122): number analyzed (Participants) | 122
  Week 48 (n=122) | -0.08 [-0.35 to 0.00]

4. Secondary Outcome: Presence of Choroidal Neovascularization (CNV) Lesion Area Measured by Optical Coherence Tomography-Angiograph (OCT-A) From Baseline to Week 48
Description: as for outcome 2
Time Frame: Baseline, Week 48
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 153
Participants
  Present CNV at baseline and Present CNV at Week 48 | 66
  Present CNV at baseline and Not Present CNV at Week 48 | 48
  Present CNV at baseline and Ungradable at Week 48 | 6
  Not Present CNV at Baseline and Present CNV at Week 48 | 5
  Not Present CNV at Baseline and Not Present CNV at Week 48 | 4
  Not Present CNV at Baseline and Ungradable at Week 48 | 1
  Ungradable at Baseline and Present CNV at Week 48 | 8
  Ungradable at Baseline and Not Present CNV at Week 48 | 14
  Ungradable at Baseline and Ungradable at Week 48 | 1
  Total at Baseline and Present CNV at Week 48 | 79
  Total at Baseline and Not Present CNV at Week 48 | 66
  Total at Baseline and Ungradable at Week 48 | 8
  Total at Baseline and Total at Week 48 | 153

5. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA) From Baseline up to Week 48
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Visual Function of the study eye was assessed using the ETDRS protocol. Participants with a BCVA ETDRS letter score of 78 to 23 (approximate Snellen equivalent of 20/32 to 20/320) in the study eye were included.
  Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
Time Frame: Baseline, Weeks 4, 8, 12, 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ETDRS letters read
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 199
ETDRS letters read
  Week 4 (n=174): number analyzed (Participants) | 174
  Week 4 (n=174) | 5.0 (7.48)
  Week 8 (n=153): number analyzed (Participants) | 153
  Week 8 (n=153) | 6.7 (8.07)
  Week 12 (n=199) | 6.7 (9.09)
  Week 48 (n=158): number analyzed (Participants) | 158
  Week 48 (n=158) | 8.3 (12.03)

6. Secondary Outcome: Percentage of Patients Who Are Maintained on an Exclusive Treatment Interval Every 12 Weeks (q12w) Following the Loading Phase to Week 48
Description: To estimate the proportion of patients treated at q12w frequency with brolucizumab.
Time Frame: Weeks 20, 32, 44, 48
Population: FAS
Measure: Number (95% Confidence Interval); unit: % of Participants
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 210
% of Participants
  % of patients with exclusive q12w dose - Week 20 | 74.5 [66.8 to 81.2]
  % of patients with exclusive q12w dose - Week 32 | 55.6 [47.3 to 63.6]
  % of patients with exclusive q12w dose - Week 44 | 42.5 [34.5 to 50.7]
  % of patients with exclusive q12w dose - Week 48 | 42.5 [34.5 to 50.7]

7. Secondary Outcome: The Probability of the First q12w Interval for Determining Successful q12w Maintenance
Description: To estimate the predictive value of the first q12w cycle for maintenance of q12w treatment with brolucizumab via the Kaplan-Meier method.
Time Frame: Weeks 0,4,5,8,9,15,16,17,18,20,21,22,24,32,33,34,35,40,41,43,44,48
Population: FAS
Measure: Number (95% Confidence Interval); unit: Probability of Q12 maintain
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 210
Probability of Q12 maintain
  Week 0 | 1 [1 to 1]
  Week 4 (n=201): number analyzed (Participants) | 201
  Week 4 (n=201) | 1 [1 to 1]
  Week 5 (n=198): number analyzed (Participants) | 198
  Week 5 (n=198) | 1 [1 to 1]
  Week 8 (n=196): number analyzed (Participants) | 196
  Week 8 (n=196) | 1 [1 to 1]
  Week 9 (n=184): number analyzed (Participants) | 184
  Week 9 (n=184) | 1 [1 to 1]
  Week 15 (n=176): number analyzed (Participants) | 176
  Week 15 (n=176) | 0.97 [0.933 to 0.988]
  Week 16 (n=171): number analyzed (Participants) | 171
  Week 16 (n=171) | 0.78 [0.716 to 0.838]
  Week 17 (n=138): number analyzed (Participants) | 138
  Week 17 (n=138) | 0.66 [0.590 to 0.729]
  Week 18 (n=117): number analyzed (Participants) | 117
  Week 18 (n=117) | 0.65 [0.572 to 0.713]
  Week 20 (n=114): number analyzed (Participants) | 114
  Week 20 (n=114) | 0.57 [0.492 to 0.638]
  Week 21 (n=97): number analyzed (Participants) | 97
  Week 21 (n=97) | 0.51 [0.433 to 0.581]
  Week 22 (n=87): number analyzed (Participants) | 87
  Week 22 (n=87) | 0.5 [0.427 to 0.575]
  Week 24 (n=86): number analyzed (Participants) | 86
  Week 24 (n=86) | 0.5 [0.422 to 0.569]
  Week 32 (n=85): number analyzed (Participants) | 85
  Week 32 (n=85) | 0.47 [0.393 to 0.540]
  Week 33 (n=80): number analyzed (Participants) | 80
  Week 33 (n=80) | 0.46 [0.382 to 0.529]
  Week 34 (n=78): number analyzed (Participants) | 78
  Week 34 (n=78) | 0.45 [0.376 to 0.523]
  Week 35 (n=77): number analyzed (Participants) | 77
  Week 35 (n=77) | 0.45 [0.376 to 0.523]
  Week 40 (n=76): number analyzed (Participants) | 76
  Week 40 (n=76) | 0.45 [0.376 to 0.523]
  Week 41 (n=72): number analyzed (Participants) | 72
  Week 41 (n=72) | 0.45 [0.376 to 0.523]
  Week 43 (n=71): number analyzed (Participants) | 71
  Week 43 (n=71) | 0.45 [0.376 to 0.523]
  Week 44 (n=65): number analyzed (Participants) | 65
  Week 44 (n=65) | 0.45 [0.376 to 0.523]
  Week 48 (n=65): number analyzed (Participants) | 65
  Week 48 (n=65) | 0.45 [0.376 to 0.523]

8. Secondary Outcome: Time From Last Intravitreal (IVT) Injection in the Initiation Phase to First Visit With no Disease Activity - Probability of no Disease Activity
Description: To evaluate the time from last IVT injection in the initiation phase to first visit with no disease activity.
  The 95% CI are estimated by using the Greenwood formula Kaplan-Meier (KM) method.
Time Frame: Week 8 until Week 41
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Probability of no disease activity
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 210
Probability of no disease activity
  Week 8 | 0.83 [0.77 to 0.88]
  Week 9 | 0.85 [0.79 to 0.90]
  Week 10 | 0.86 [0.80 to 0.91]
  Week 15 | 0.86 [0.80 to 0.91]
  Week 16 | 0.87 [0.81 to 0.92]
  Week 18 | 0.88 [0.82 to 0.93]
  Week 23 | 0.89 [0.83 to 0.94]
  Week 24 | 0.9 [0.84 to 0.95]
  Week 31 | 0.9 [0.84 to 0.95]
  Week 32 | 0.93 [0.87 to 0.97]
  Week 33 | 0.94 [0.88 to 0.98]
  Week 35 | 0.96 [0.90 to 0.99]
  Week 36 | 0.96 [0.90 to 0.99]
  Week 41 | 0.96 [0.90 to 0.99]

9. Secondary Outcome: Change From Baseline up to Week 48 in SD-OCT Assessed by Qualitative and Quantitative Criteria: Central Sub-Field Retinal Thickness (CSFT)
Description: Central sub-field thickness (CSFT) was measured by Spectral Domain Optical Coherence Tomography (SD-OCT). The CSFT evaluated in this study represents the average retinal thickness of the circular area within 1 mm diameter around the foveal center. SD-OCT images were obtained and assessed in the study eye by SD-OCT machines. (i.e. no time-domain nor swept-source OCT).
Time Frame: Baseline, Weeks 4, 8, 12, 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 188
μm
  Week 4 (n=164): number analyzed (Participants) | 164
  Week 4 (n=164) | -131.79 (109.100)
  Week 8 (n=143): number analyzed (Participants) | 143
  Week 8 (n=143) | -152.95 (128.031)
  Week 12 (n=188) | -150.51 (126.931)
  Week 48 (n=150): number analyzed (Participants) | 150
  Week 48 (n=150) | -151.09 (134.684)

10. Secondary Outcome: Change From Baseline up to Week 48 in SD-OCT and FA Features Assessed by Qualitative and Quantitative Criteria: Sub and Intraretinal Fluid, Sub-RPE (Retinal Pigmented Epithelium) - Study Eye
Description: To evaluate the effect of brolucizumab on anatomical parameters as assessed by Spectral Domain Optical Coherence Tomography (SD-OCT) and Fluorescein Angiography (FA).
  RPE = Retinal Pigmented Epithelium IRF = Intraretinal Fluid SRF = Subretinal Fluid Sub-RPE = Sub Retinal Pigmented Epithelium
Time Frame: Baseline, Weeks 4, 8, 12, 48
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 201
Participants
  Baseline Intraretinal fluid | 101
  Baseline Subretinal fluid | 169
  Baseline Sub-RPE fluid | 60
  Baseline Without any fluid (IRF/SRF) | 8
  Baseline With any fluid (IRF/SRF) | 193
  Week 4 Intraretinal fluid (n=174 ): number analyzed (Participants) | 174
  Week 4 Intraretinal fluid (n=174 ) | 39
  Week 4 Subretinal fluid (n=174 ): number analyzed (Participants) | 174
  Week 4 Subretinal fluid (n=174 ) | 69
  Week 4 Sub-RPE fluid (n=174 ): number analyzed (Participants) | 174
  Week 4 Sub-RPE fluid (n=174 ) | 47
  Week 4 Without any fluid (IRF/SRF) (n=174 ): number analyzed (Participants) | 174
  Week 4 Without any fluid (IRF/SRF) (n=174 ) | 84
  Week 4 With any fluid (IRF/SRF) (n=174 ): number analyzed (Participants) | 174
  Week 4 With any fluid (IRF/SRF) (n=174 ) | 90
  Week 8 Intraretinal fluid (n=155): number analyzed (Participants) | 155
  Week 8 Intraretinal fluid (n=155) | 31
  Week 8 Subretinal fluid (n=155): number analyzed (Participants) | 155
  Week 8 Subretinal fluid (n=155) | 28
  Week 8 Sub-RPE fluid (n=155): number analyzed (Participants) | 155
  Week 8 Sub-RPE fluid (n=155) | 50
  Week 8 Without any fluid (IRF/SRF) (n=155): number analyzed (Participants) | 155
  Week 8 Without any fluid (IRF/SRF) (n=155) | 108
  Week 8 With any fluid (IRF/SRF) (n=155): number analyzed (Participants) | 155
  Week 8 With any fluid (IRF/SRF) (n=155) | 44
  Week 12 Intraretinal fluid (n=197): number analyzed (Participants) | 197
  Week 12 Intraretinal fluid (n=197) | 51
  Week 12 Subretinal fluid (n=197): number analyzed (Participants) | 197
  Week 12 Subretinal fluid (n=197) | 38
  Week 12 Sub-RPE fluid (n=197): number analyzed (Participants) | 197
  Week 12 Sub-RPE fluid (n=197) | 19
  Week 12 Without any fluid (IRF/SRF) (n=197): number analyzed (Participants) | 197
  Week 12 Without any fluid (IRF/SRF) (n=197) | 120
  Week 12 With any fluid (IRF/SRF) (n=197): number analyzed (Participants) | 197
  Week 12 With any fluid (IRF/SRF) (n=197) | 74
  Week 48 Intraretinal fluid (n=159): number analyzed (Participants) | 159
  Week 48 Intraretinal fluid (n=159) | 38
  Week 48 Subretinal fluid (n=159): number analyzed (Participants) | 159
  Week 48 Subretinal fluid (n=159) | 26
  Week 48 Sub-RPE fluid (n=159): number analyzed (Participants) | 159
  Week 48 Sub-RPE fluid (n=159) | 19
  Week 48 Without any fluid (IRF/SRF) (n=159): number analyzed (Participants) | 159
  Week 48 Without any fluid (IRF/SRF) (n=159) | 99
  Week 48 With any fluid (IRF/SRF) (n=159): number analyzed (Participants) | 159
  Week 48 With any fluid (IRF/SRF) (n=159) | 60

11. Secondary Outcome: Incidence of Adverse Events (AEs) (Serious and Nonserious) Reported in Patients Treated With Brolucizumab.
Description: An AE is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study.
Time Frame: Up to Week 48
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 210
Participants
  Any Adverse Event (AE) - Ocular | 95
  Any AE - Treatment-related - Ocular | 32
  Any AE - Procedure-related - Ocular | 18
  Serious Adverse events (SAE) - Ocular | 8
  SAEs - Treatment-related - Ocular | 7
  SAEs - Procedure-related -Ocular | 1
  Fatal SAEs - Ocular | 0
  Fatal SAEs - Treatment-related - Ocular | 0
  Fatal SAEs - Procedure-related - Ocular | 0
  AEs leading to treatment discontinuation - Ocular | 25
  AEs leading to treatment disc - Treatment-related - Ocular | 25
  AEs leading to treatment disc - Procedure-related - Ocular | 6
  AEs leading to interruption - Ocular | 0
  AEs leading to interruption -Treatment-related - Ocular | 0
  AEs leading to interruption - Procedure-related - Ocular | 0
  Any Adverse Event - Non-Ocular | 77
  Any AE - Treatment-related - Non-Ocular | 1
  Any AE - Procedure-related - Non-Ocular | 0
  Serious Adverse events (SAE) - Non-Ocular | 13
  SAEs - Treatment-related - Non-Ocular | 0
  SAEs - Procedure-related - Non-Ocular | 0
  Fatal SAEs - Non-Ocular | 1
  Fatal SAEs - Treatment-related - Non-Ocular | 0
  Fatal SAEs - Procedure-related - Non-Ocular | 0
  AEs leading to treatment discontinuation - Non-Ocular | 3
  AEs leading to treatment disc - Treatment-related - Non-Ocular | 1
  AEs leading to treatment disc - Procedure-related - Non-Ocular | 0
  AEs leading to interruption - Non-Ocular | 0
  AEs leading to interruption - Treatment-related - Non-Ocular | 0
  AEs leading to interruption - Procedure-related - Non-Ocular | 0
  Any Adverse Event - All patients | 135
  Any AE - Treatment-related - All patients | 33
  Any AE - Procedure-related All patients | 18
  Serious Adverse events (SAE) - All patients | 20
  SAEs - Treatment-related - All patients | 7
  SAEs - Procedure-related - All patients | 1
  Fatal SAEs - All patients | 1
  Fatal SAEs - Treatment-related - All patients | 0
  Fatal SAEs - Procedure-related - All patients | 0
  AEs leading to treatment discontinuation - All patients | 28
  AEs leading to treatment disc - Treatment-related - All patients | 26
  AEs leading to treatment disc - Procedure-related - All patients | 6
  AEs leading to interruption - All patients | 0
  AEs leading to interruption - Treatment-related - All patients | 0
  AEs leading to interruption - Procedure-related - All patients | 0

12. Secondary Outcome: Incidence of AEs (Serious and Nonserious) Reported in Patients Treated With Brolucizumab, by Primary System Organ Class (SOC) and Preferred Term (PT) - Ocular Adverse Events in Study Eye
Description: as for outcome 11
Time Frame: Up to Week 48
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 210
Participants
  Number of patients with at least one AE | 85
  Eye disorders | 81
  - Eye pain | 10
  - Vitritis | 10
  - Dry eye | 9
  - Vitreous floaters | 8
  - Vision blurred | 6
  - Visual acuity reduced | 6
  - Cataract | 5
  - Ocular hypertension | 5
  - Retinal haemorrhage | 5
  - Uveitis | 5
  - Keratitis | 4
  - Conjunctival haemorrhage | 3
  - Eye pruritus | 3
  - Iridocyclitis | 3
  -Lacrimation increased | 3
  - Retinal pigment epithelial tear | 3
  - Retinal vasculitis | 3
  - Vitreous detachment | 3
  - Blepharitis | 2
  - Metamorphopsia | 2
  - Ocular discomfort | 2
  - Ocular vasculitis | 2
  - Photophobia | 2
  - Punctate keratitis | 2
  - Retinal degeneration | 2
  - Retinal occlusive vasculitis | 2
  - Serous retinal detachment | 2
  - Visual field defect | 2
  - Anterior chamber cell | 1
  - Anterior chamber inflammation | 1
  - Conjunctivitis allergic | 1
  - Detachment of macular retinal pigment epithelium | 1
  - Diplopia | 1
  - Eye inflammation | 1
  - Eye irritation | 1
  - Foreign body sensation in eyes | 1
  - Ocular hyperaemia | 1
  - Periorbital pain | 1
  - Photopsia | 1
  - Posterior capsule opacification | 1
  - Retinal fibrosis | 1
  - Retinal neovascularisation | 1
  - Retinal oedema | 1
  - Retinal perivascular sheathing | 1
  - Vitreoretinal traction syndrome | 1
  - Vitreous haze | 1
  Immune system disorders | 2
  - Drug hypersensitivity | 1
  - Seasonal allergy | 1
  Infections and infestations | 1
  - Conjunctivitis | 1
  Injury, poisoning and procedural complications | 3
  - Foreign body in eye | 1
  - Postoperative hypertension | 1
  - Procedural pain | 1
  Investigations | 1
  - Intraocular pressure increased | 1

13. Secondary Outcome: Incidence of AEs (Serious and Nonserious) Reported in Patients Treated With Brolucizumab - Non-Ocular Adverse Events
Description: as for outcome 11
Time Frame: Up to Week 48
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | RTH258/Brolucizumab
Number analyzed (Participants) | 210
Participants | 77

ADVERSE EVENTS:
Time Frame: Adverse events are reported from first dose of study treatment plus 30 days post treatment (if last treatment was at Week 40) or 60 days post treatment (if last dose was at Week 44), for a maximum reporting period of 48 weeks.
Arm/Group | RTH258/Brolucizumab
All-Cause Mortality (participants affected / at risk) | 1/210
Serious Adverse Events (participants affected / at risk) | 20/210
Other Adverse Events (participants affected / at risk) | 130/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RTH258/Brolucizumab (N=210)
Aortic valve incompetence (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Eye haematoma - Fellow eye (Eye disorders) | 1
Iridocyclitis - Study eye (Eye disorders) | 1
Uveitis - Study eye (Eye disorders) | 3
Vitritis - Study eye (Eye disorders) | 4
Autoimmune pancreatitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Aortic dissection (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Peripheral artery stenosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RTH258/Brolucizumab (N=210)
Anaemia (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Age-related macular degeneration - Fellow eye (Eye disorders) | 1
Anterior chamber cell - Study eye (Eye disorders) | 1
Anterior chamber inflammation - Study eye (Eye disorders) | 1
Blepharitis (Eye disorders) | 3
Blepharitis - Both eye (Eye disorders) | 2
Cataract - Both eye (Eye disorders) | 2
Cataract - Fellow eye (Eye disorders) | 2
Cataract - Study eye (Eye disorders) | 3
Chalazion (Eye disorders) | 3
Conjunctival haemorrhage - Both eye (Eye disorders) | 1
Conjunctival haemorrhage - Study eye (Eye disorders) | 2
Conjunctivitis allergic - Both eye (Eye disorders) | 1
Detachment of macular retinal pigment epithelium - Study eye (Eye disorders) | 1
Detachment of retinal pigment epithelium - Fellow eye (Eye disorders) | 1
Diplopia - Both eye (Eye disorders) | 1
Dry eye - Both eye (Eye disorders) | 7
Dry eye - Study eye (Eye disorders) | 2
Eye inflammation - Study eye (Eye disorders) | 1
Eye irritation - Study eye (Eye disorders) | 1
Eye pain - Both eye (Eye disorders) | 2
Eye pain - Fellow eye (Eye disorders) | 1
Eye pain - Study eye (Eye disorders) | 8
Eye pruritus - Both eye (Eye disorders) | 1
Eye pruritus - Study eye (Eye disorders) | 2
Eyelid ptosis (Eye disorders) | 1
Eyelids pruritus (Eye disorders) | 1
Foreign body sensation in eyes - Both eye (Eye disorders) | 1
Foreign body sensation in eyes - Study eye (Eye disorders) | 1
Iridocyclitis - Study eye (Eye disorders) | 2
Keratitis - Both eye (Eye disorders) | 2
Keratitis - Fellow eye (Eye disorders) | 2
Keratitis - Study eye (Eye disorders) | 2
Lacrimation increased - Both eye (Eye disorders) | 1
Lacrimation increased - Fellow eye (Eye disorders) | 1
Lacrimation increased - Study eye (Eye disorders) | 2
Metamorphopsia - Study eye (Eye disorders) | 2
Neovascular age-related macular degeneration - Fellow eye (Eye disorders) | 10
Ocular discomfort - Study eye (Eye disorders) | 2
Ocular hyperaemia - Study eye (Eye disorders) | 1
Ocular hypertension - Both eye (Eye disorders) | 1
Ocular hypertension - Study eye (Eye disorders) | 4
Ocular vasculitis - Study eye (Eye disorders) | 2
Periorbital pain - Both eye (Eye disorders) | 1
Photophobia - Both eye (Eye disorders) | 1
Photophobia - Study eye (Eye disorders) | 1
Photopsia - Both eye (Eye disorders) | 1
Posterior capsule opacification - Both eye (Eye disorders) | 1
Posterior capsule opacification - Fellow eye (Eye disorders) | 1
Punctate keratitis - Study eye (Eye disorders) | 2
Retinal cyst - Fellow eye (Eye disorders) | 1
Retinal degeneration - Study eye (Eye disorders) | 2
Retinal fibrosis - Study eye (Eye disorders) | 1
Retinal haemorrhage - Both eye (Eye disorders) | 2
Retinal haemorrhage - Study eye (Eye disorders) | 3
Retinal neovascularisation - Study eye (Eye disorders) | 1
Retinal occlusive vasculitis - Study eye (Eye disorders) | 2
Retinal oedema - Study eye (Eye disorders) | 1
Retinal perivascular sheathing - Study eye (Eye disorders) | 1
Retinal pigment epithelial tear - Study eye (Eye disorders) | 3
Retinal vasculitis - Study eye (Eye disorders) | 3
Serous retinal detachment - Fellow eye (Eye disorders) | 2
Serous retinal detachment - Study eye (Eye disorders) | 2
Swelling of eyelid (Eye disorders) | 1
Uveitis - Study eye (Eye disorders) | 2
Vision blurred - Both eye (Eye disorders) | 1
Vision blurred - Study eye (Eye disorders) | 5
Visual acuity reduced - Both eye (Eye disorders) | 1
Visual acuity reduced - Study eye (Eye disorders) | 5
Visual field defect - Fellow eye (Eye disorders) | 1
Visual field defect - Study eye (Eye disorders) | 2
Vitreoretinal traction syndrome - Study eye (Eye disorders) | 1
Vitreous detachment - Study eye (Eye disorders) | 3
Vitreous floaters - Both eye (Eye disorders) | 1
Vitreous floaters - Fellow eye (Eye disorders) | 2
Vitreous floaters - Study eye (Eye disorders) | 8
Vitreous haze - Study eye (Eye disorders) | 1
Vitritis - Study eye (Eye disorders) | 6
Aerophagia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 2
Dental cyst (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 2
Cholestasis (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Drug hypersensitivity - Both eye (Immune system disorders) | 1
Seasonal allergy - Both eye (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 2
COVID-19 (Infections and infestations) | 8
Conjunctivitis - Fellow eye (Infections and infestations) | 1
Conjunctivitis - Study eye (Infections and infestations) | 1
Conjunctivitis viral - Fellow eye (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Arthropod bite (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Foreign body in eye - Study eye (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 2
Joint injury (Injury, poisoning and procedural complications) | 2
Lip injury (Injury, poisoning and procedural complications) | 1
Postoperative hypertension - Study eye (Injury, poisoning and procedural complications) | 1
Procedural pain - Study eye (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2
Blood cholesterol increased (Investigations) | 1
Intraocular pressure increased - Study eye (Investigations) | 1
SARS-CoV-2 test positive (Investigations) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Balance disorder (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 3
Ischaemic stroke (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Retinal migraine (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
White matter lesion (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT04239027/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/27/NCT04239027/SAP_001.pdf